CLINICAL TRIAL: NCT01245231
Title: Stat3 Activation as a Potential Prognostic Marker and Therapeutic Target in Pediatric AML-II
Brief Title: Prognostic Biomarkers in Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B6; COG-AAML11B6 (Other: Children's Oncology Group); CDR0000689410 (Other: Clinical Trials.gov); NCI-2011-02845 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Blotting, Western; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: protein expression analysis
Genetic: western blotting
Other: flow cytometry
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood or tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is studying prognostic biomarkers in cell samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the percentage of primary acute myeloid leukemia (AML) samples with increased Stat3 signaling pathway activity.
* To evaluate the presence of constitutive Stat3 activation and the sensitivity of Stat3 activation to low- and high-doses of cytokines.
* To evaluate the expression levels of Stat3 protein and the upstream and downstream regulators of Stat3 activation.

Secondary

* To classify samples according to a Stat3 activation pattern and correlate this result with event-free survival (EFS) and overall survival (OS).

OUTLINE: Cryopreserved AML specimens are analyzed for pStat3 and pStat5 levels, response to cytokine levels, and expression level of proteins known to influence stat activity by flow cytometry and western blot assays. Results are also compared with prognostic variables determined in CCG-291 study, including age, race, WBC, and cytogenetic risks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)
* Cryopreserved AML specimens

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of acute myeloid leukemia (AML)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-05; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Correlation of constitutive pStat3 with inducible pStat3
Correlation of pStat3 responses with pStat5 responses, and G-CSF-induced responses with IL-6- induced responses
Correlation of pStat3- and pStat5-induced responses with surface G-CSFR and gp130 expression
Correlation of constitutive pStat3/pStat5 with levels of the negative regulators SOCS3 and SHP1

SECONDARY OUTCOMES:
Correlation between pStat3/pStat5 and event-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Michele S. Redell, MD, PhD, Principal Investigator — Texas Children's Cancer Center